CLINICAL TRIAL: NCT01480219
Title: Evaluation Of The Importance Of Risk-Factor Adjustment For Assessing The Relationship Between Voriconazole Utilization And The Development Of Non-Melanoma Skin Cancer Among Lung And Heart/Lung Transplant Patients, 2002-2009
Brief Title: Evaluation Of The Importance Of Risk-Factor Adjustment For Assessing The Relationship Between Voriconazole Utilization And The Development Of Non-Melanoma Skin Cancer Among Lung And Heart/Lung Transplant Patients, 2002-2009g
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: A1501098
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Results first posted 2013-03-11 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-02

CONDITIONS: Non-Melanoma Skin Carcinoma
Keywords: voriconazole; non-melanoma skin cancer; confounding; statistical adjustment; risk adjustment; lung transplant; heart/lung transplant; immunosuppression
MeSH Terms: interventions — Voriconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Any Voriconazole
  Interventions: Drug: voriconazole (Vfend)
- No Voriconazole
  Interventions: Other: no voriconazole (Vfend)

INTERVENTIONS:
Drug: voriconazole (Vfend) — Voriconazole utilization was identified as any vs. none for the period 180 days before and 180 days after the date of transplant.
  Other Names: Vfend
  Groups: Any Voriconazole
Other: no voriconazole (Vfend) — Voriconazole utilization was identified as any vs. none for the period 180 days before and 180 days after the date of transplant.
  Other Names: Vfend
  Groups: No Voriconazole

SUMMARY:
The primary objective of the study is to assess the relationship (both crude and adjusted) between voriconazole utilization and the development of non-melanoma skin cancer among adult patients who received a lung or heart/lung transplant and were continuously enrolled in a large U.S. commercial health plan.

DETAILED DESCRIPTION:
N/A. All patients aged 18 or older who received a lung or heart/lung transplant from January 1, 2002 through December 31, 2009 in the MarketScan database were sampled.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older who received a lung or heart/lung transplant from January 1, 2002 through December 31, 2009 in the MarketScan database will be initially included in the study.

Exclusion Criteria:

* Patients who are younger than 18 years of age and who are not enrolled for at least 180 days before and 180 days after the date of transplant will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or older who received a lung or heart/lung transplant from January 1, 2002 through December 31, 2009 in the MarketScan database will be initially included in the study. Patients who are younger than 18 years of age and who are not enrolled for at least 180 days before and 180 days after the date of transplant will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501098&StudyName=Evaluation%20Of%20The%20Importance%20Of%20Risk-Factor%20Adjustment%20For%20Assessing%20The%20Relationship%20Between%20Voriconazole%20Utilization%20And%20The%20Development%20O

RESULTS

PARTICIPANT FLOW:
Groups:
- No Voriconazole: Participants not having any voriconazole prescription claims in the period 180 days before or after the date of lung or heart/lung transplant.
- Voriconazole: Participants having any voriconazole prescription claims in the period 180 days before or after the date of lung or heart/lung transplant.
Period: Overall Study
Arm/Group | No Voriconazole | Voriconazole
Started | 325 | 142
Completed | 325 | 142
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Voriconazole | Voriconazole | Total
Number analyzed (Participants) | 325 | 142 | 467
Age, Customized [Number; unit: participants]
  18 to 29 years | 20 | 10 | 30
  30 to 49 years | 65 | 22 | 87
  50 to 59 years | 105 | 44 | 149
  60 to 69 years | 121 | 60 | 181
  Greater than or equal to 70 years | 14 | 6 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 47 | 189
  Male | 183 | 95 | 278

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Non-Melanoma Skin Cancer (NMSC)
Time Frame: Baseline until non-melanoma skin cancer diagnosis, loss-to-follow-up due to death or termination of the health plan or end of the study, assessed up to Year 8
Population: Final analysis set included participants who met the eligibility criteria.
Measure: Number; unit: participants
Arm/Group | No Voriconazole | Voriconazole
Number analyzed (Participants) | 325 | 142
participants | 34 | 23
Statistical Analysis 1: Comparison: No Voriconazole vs Voriconazole; Crude hazard ratio (HR) and corresponding 95 percent (%) confidence interval (CI) were calculated using an unadjusted Cox proportional hazards regression model; Test type: Superiority or Other; p = 0.042, Regression, Cox; Hazard Ratio (HR) = 1.74, 95% CI 2-sided [1.02 to 2.96]
Statistical Analysis 2: Comparison: No Voriconazole vs Voriconazole; HR and corresponding 95% CI were calculated using a parsimoniously adjusted Cox proportional hazards regression model; Test type: Superiority or Other; p = 0.453, Regression, Cox; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.71 to 2.14]

ADVERSE EVENTS:
Description: Safety data was not collected as this was a retrospective study.
Arm/Group | No Voriconazole | Voriconazole
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.